| 1 | Clinical Efficacy of Cefixime for Treatment of Early Syphilis |
|---|---------------------------------------------------------------|
| 2 | NCT:03660488 |
| 3 | August 10, 2020 |

# 4 Clinical Trial Protocol to Evaluate the Efficacy of Cefixime in the

5 Treatment of Early Syphilis

6 7

- 8 Authors: SN Mehta<sup>1</sup>, C. Stafylis<sup>1</sup>, D. Tellalian<sup>2</sup>, P. Burian<sup>2</sup>, C. Okada<sup>2</sup>, C. Millner<sup>2</sup>, C. Mejia<sup>3</sup> JD
- 9 Klausner<sup>1,2</sup>

10

11

#### Abstract

- 12 **Background:** Syphilis rates have been increasing both in the US and internationally with
- incidence higher among men-who-have-sex-with-men and people living with human
- immunodeficiency virus (HIV) infection. Currently, benzathine penicillin is the recommended
- treatment for syphilis in all patients. Global shortages and cost increases in benzathine penicillin
- call for alternative treatment options. This study evaluates the efficacy of oral cefixime for the
- 17 treatment of early syphilis.
- 18 **Methods:** We are conducting a randomized, multisite, open-label, non-comparative clinical trial
- in Los Angeles and Oakland, California. Eligible participants are >18 years old, with primary,
- secondary or early latent syphilis (Rapid Plasma Reagin [RPR] titer ≥1:8). Patients with HIV
- infection must have a viral load  $\leq 200$  copies/mL and CD4+ T cell count  $\geq 350$  cells/ $\mu$ l during the
- 22 past 6 months. Participants are randomized to receive either 2.4M IU benzathine penicillin G
- 23 intramuscularly once or cefixime 400mg orally twice a day for 10 days. Participants return at 3, 6,
- 24 and 12 months post-treatment for follow-up RPR serological testing. The primary outcome is the
- proportion of participants who achieve ≥4-fold RPR titer decrease at 3- or 6-months post-
- 26 treatment.
- 27 **Discussion:** Clinical trials evaluating the efficacy of alternative antibiotics to penicillin are urgently
- 28 needed.
- 29 Trial Registration: Clinicaltrials.gov, NCT03660488. Registered September 4, 2018,

31

32

30

# Keywords

33 Clinical Trial, Cefixime, *Treponema pallidum*, penicillin, early syphilis, syphilis

34

35

## **Administrative information**

37

36

| Title {1} | Clinical Trial Evaluating the Clinical Efficacy of Cefixime in Treatment for Early Syphilis |
|---|---|
| Trial registration {2a and 2b}. | ClinicalTrials.gov Identifier: NCT03660488 (1) |
| Protocol version {3} | Version 9; 11.20.2019 |
| Funding {4} | AIDS Healthcare Foundation research grant (Grant #20181796) |
| Author details {5a} | <ol> <li>Department of Medicine, David Geffen School of Medicine at UCLA, Los Angeles, CA/United States of America</li> <li>Department of Medicine, AIDS Healthcare Foundation, Los Angeles, CA/United States of America</li> <li>Public Health Division, AIDS Healthcare Foundation, Los Angeles, CA/United States of America</li> </ol> |
| Name and contact information for the trial sponsor {5b} | AIDS Healthcare Foundation |

| Role of sponsor {5c} | The sponsor played no part in study design; and will play no part in the collection, management, analysis, and interpretation of data; writing of the |
|---|---|
| | report; and the decision to submit the report for publication. |

#### Introduction

39

63

40 **Background and rationale {6a}** Syphilis rates have been increasing both in the US and internationally, with incidence higher among 41 42 men-who-have-sex-with-men and people living with human immunodeficiency virus (HIV) 43 infection (2-4). Currently, benzathine penicillin is the recommended treatment for syphilis in all 44 patients, including those living with HIV infection. Doxycycline and tetracycline are available 45 alternative treatments for non-pregnant patients who are allergic to penicillin (5-8). Injectable daily 46 ceftriaxone is another alternative treatment that may be considered and is safe in pregnancy, as a 47 recent review from our team showed (9). 48 Existing alternative treatment recommendations are based on clinical experience, a limited number 49 of small clinical trials, and case series (5-7, 10). However, each regimen poses clinical challenges. 50 Doxycycline/tetracycline require 14 days of treatment by mouth, with tetracycline requiring four 51 daily doses. Ceftriaxone is administered intramuscularly, just like penicillin, but it requires daily 52 injections for 10-14 days, making adherence potentially problematic. In pregnancy, only benzathine 53 penicillin is recommended due to potential toxic effects of the alternatives or due to insufficient 54 efficacy data (WHO). Shortages of benzathine penicillin worldwide have led to the use of unproven 55 non-penicillin alternatives (10-12). Considering the high cost and time required for developing and approving new antibiotics that can 56 57 treat syphilis in patients with and without HIV infection, a new approach for identifying new, safe, 58 and efficacious antibiotic treatments for syphilis is necessary. Previously Food and Drug 59 Administration (FDA)-approved antibiotics, that are safe and efficacious in other infections and have 60 a favorable pharmacologic profile suggesting activity against *Treponema pallidum*, may be effective 61 alternatives for treating syphilis. 62 Cefixime is an FDA-approved orally administered third-generation cephalosporin with spectrum of

activity and pharmacokinetic profile similar to that of ceftriaxone, a drug which has been used for the

64 treatment for syphilis (13). Cefixime is clinically used for uncomplicated urinary tract infections, 65 upper respiratory tract bacterial infections and in the treatment of uncomplicated Neisseria gonorrhoeae genital infection (14). To our knowledge, it has never been studied as a treatment for 66 67 early syphilis. 68 Cefixime has a well-studied pharmacokinetic profile (14-19). Unlike other alternatives for syphilis, 69 adverse event profiles are favorable with cefixime in non-pregnant as well as pregnant patients (20, 70 21). Nearly 40-50% of the dose is absorbed when it is given orally, whether administered with or 71 without food. Peak concentrations occur between 2 and 6 hours following oral administration of a 72 single 400mg tablet. A single 400mg tablet produces an average peak concentration of approximately 73 3.7µg/mL (range 1.3-7.7µg/mL). Typical blood levels of cefixime after a single dose of cefixime 400 74 mg by mouth are 4.84 µg/ml maximum at 4 hours and above 1.0 µg/ml at 12 hours. Serum protein 75 binding is concentration independent with a bound fraction of approximately 65%. Cefixime is 76 moderately distributed into extracellular water/tissue pools. Its half-life averages to 3-4 hours but 77 may range up to 9 hours in healthy volunteers. Approximately 50% of the absorbed dose is excreted 78 unmodified in the urine within 24 hours and nearly 10% is excreted in bile (10). 79 We therefore believe that cefixime's pharmacokinetic similarity to ceftriaxone and its safety in the 80 treatment of pregnant women could potentially make it a viable option in the treatment of early

82

83

84

85

86

81

#### Objective {7}

syphilis.

The primary objective of our study is to determine the efficacy of cefixime 400mg, taken orally two times a day (BID) for 10 consecutive days. Our hypothesis is that cefixime would be an efficacious treatment for early syphilis.

87

88

## Trial design {8}

| 89 | This is a randomized, open-label, non-comparative pilot clinical trial. Participants will be randomly |
|---|---|
| 90 | assigned (1:1 allocation) to receive either the standard of care benzathine penicillin injection or 10- |
| 91 | days of oral cefixime. The study will require 2 years to be completed and each participant will be part |
| 92 | of the study for one year. |
| 93 | |
| 94 | Methods: Participants, interventions and outcomes |
| 95 | Study setting {9} |
| 96 | The study will take place in 3 primary care HIV healthcare clinics and 1 wellness center of the |
| 97 | AIDS Healthcare Foundation in Los Angeles and Oakland, California. Healthcare clinics offer HIV |
| 98 | and sexually transmitted infection (STI) primary care services while wellness centers are walk-in |
| 99 | comprehensive sexual health clinics that offer HIV/STI screening services, STI treatment and other |
| 100 | prevention services. |
| 101 | |
| 102 | Eligibility criteria {10} |
| 103 | The inclusion criteria are: |
| 104 | 1) Clinically or laboratory confirmed new cases of early syphilis (primary, secondary, early |
| 105 | latent syphilis) with a plasma Rapid Plasma Reagin (RPR) ≥ 1:8 |
| 106 | 2) 18 years of age or older, capable of providing informed consent |
| 107 | 3) HIV infected individuals must have CD4 T cll count≥350 cells/mm³ and be virologically |
| 108 | suppressed (viral load < 200 copies/mL) during the past 6 months |
| 109 | 4) Able to travel to clinic once a day or be available for phone calls or receive text message for |
| 110 | at least 7-10 days |
| 111 | The exclusion criteria are: |
| 112 | 1) Allergy to cefixime or penicillin |
| 113 | 2) Pregnancy or a positive pregnancy test |

| 114 | 3) Serofast RPR fifer (prior fifer ≥1:8 without history of 4-fold fifer decline) |
|---|---|
| 115 | 4) Recent (within the past 7 days) or concomitant antimicrobial therapy with activity against |
| 116 | syphilis, namely azithromycin, doxycycline, ceftriaxone or other beta lactam antibiotics (e.g. |
| 117 | amoxicillin) |
| 118 | 5) A medical condition or other factor that might affect their ability to follow the protocol |
| 119 | |
| 120 | Who will take informed consent? {26a} |
| 121 | Patients must provide written, informed consent before any study procedures occur (randomization, |
| 122 | blood sample collection, treatment). Consent will be obtained by a study team member in a private |
| 123 | examination room. |
| 124 | |
| 125 | Additional consent provisions for collection and use of participant data and biological |
| 126 | specimens {26b} |
| 127 | Patients will also sign a Health Insurance Portability and Accountability Act (HIPAA) release form |
| 128 | allowing access to clinical and laboratory data, including their HIV test results. |
| 129 | |
| 130 | Interventions |
| 131 | Explanation for the choice of comparators {6b} |
| 132 | This is a pilot, non-comparative clinical trial designed to collect preliminary efficacy data. It |
| 133 | includes an "experimental arm" of participants receiving cefixime and a contemporaneous "control |
| 134 | arm" of participants receiving benzathine penicillin. The study was not designed to be adequately |
| 135 | powered to show a statistically significant difference in the efficacy between the penicillin and |
| 136 | cefixime arms. |
| 137 | |
| 138 | Intervention description {11a} |

Eligible participants who provide their consent are randomized to the two arms of the study. Initially, the study team collects demographic (age, gender, race, ethnicity, contact, sexual orientation) and clinical information (most recent RPR titer, CD4 T cell count, HIV viral load). A venipuncture blood sample is collected by trained clinic staff and it is sent to the laboratory for testing. Testing is conducted on serum using the Arlington scientific RPR test kit (Arlington, Virginia) (22). Participants are randomly assigned to the two treatment groups. Participants assigned to the penicillin arm will receive 1 dose of 2.4M IU benzathine penicillin G on the day of enrollment. Participants who are assigned to the cefixime arm will be given 20 capsules of oral cefixime 400mg on the day of enrollment to take for the following 10 days. Study staff observed receipt of the first dose. Subjects in the cefixime arm will then be asked to return for a clinical assessment or have a phone call assessment with the study team member 2 weeks following enrolment. Study staff will follow up with all participants at 3, 6, and 12 months. In each follow up, participants are asked questions regarding symptoms, antibiotic use in the past 3 months and number of sex partners with whom they had condom-less sex in the past 3 months. A new venipuncture blood sample is also collected for RPR testing Criteria for discontinuing or modifying allocated interventions {11b} Participants may request to leave the study or they may be withdrawn due to study-related adverse

Participants may request to leave the study or they may be withdrawn due to study-related adverse events. If a subject is discontinued from study participation due to an adverse event, they will be evaluated by the study clinicians for the need of additional treatment for syphilis. Safety data will be collected on any subject who is withdrawn from the study.

Participants in both study groups may receive additional treatment with penicillin, if they show no response to treatment (stable or absence of 4-fold decline at 6 months).

163

162

139

140

141

142

143

144

145

146

147

148

149

150

151

152

153

154

155

156

157

158

159

160

161

| 164 | Strategies to improve adherence to interventions {11c} |
|---|---|
| 165 | To ensure retention of participants, follow-up visits will be scheduled to coincide with routine clinic |
| 166 | appointments for HIV care or preventive sexual health appointments, which occur every three |
| 167 | months. In addition, study staff will contact participants, either over the phone or via text message, |
| 168 | before their scheduled follow-up appointment. Finally, participants will receive reimbursement for |
| 169 | their time and transportation in the form of a gift card. |
| 170 | |
| 171 | Relevant concomitant care permitted or prohibited during the trial {11d} |
| 172 | Usual HIV care and treatment for the participant will continue throughout the trial. Concomitant |
| 173 | antibiotic use during the participation in the study duration of the trial will be recorded. |
| 174 | |
| 175 | Provisions for post-trial care {30} |
| 176 | Once participants complete the study, they will be able to continue receiving clinical care from the |
| 177 | clinics. Participants study records will be reviewed and if necessary, additional treatment for |
| 178 | syphilis will be administered according to the standard of care protocol. |
| 179 | |
| 180 | Outcomes {12} |
| 181 | The primary outcome is the successful treatment of early syphilis by the 3-, or 6-month follow-up. |
| 182 | The participants' RPR titer will be used as the primary measure of outcome. Successful treatment is |
| 183 | defined as an equal or greater than 4-fold RPR titer decrease, from baseline to 3 or 6 months after |
| 184 | treatment. |
| 185 | |
| 186 | Participant timeline {13} |
| 187 | Participants will be part of the study for 12 months. Study evaluations will occur at 3, 6- and 12- |
| 188 | months post-treatment. See Figure 1 for the participant timeline for the trial. |
| 189 | |

#### Figure 1: Participant Enrollment and Follow-Up Schedule



## **Sample size {14}**

The primary analysis will compute the proportion of subjects with a 4-fold decrease (from study entry RPR) in RPR titer from baseline at 6 months in the per protocol analysis population. If we assume a sample size of 40 and the proportion of subjects with a 4-fold decrease in RPR from baseline at 6 months to be 0.9 (90%), we would have a 95% confidence interval of (0.76, 0.97). To calculate the number of subjects required to enroll to reach 40 evaluable subjects in the PP analysis population, the assumptions that 20% of subjects will be excluded from the PP analysis population (due to loss to follow-up or non-compliance with study medication schedule). Under that assumption, enrolling 50 subjects will provide 40 subjects in the PP analysis population.

#### **Recruitment {15}**

Participant recruitment will occur in 4 AIDS Healthcare Foundation (AHF) Clinics based in Los Angeles, California and Oakland, California. Study clinicians will review the medical and laboratory records of syphilis cases returning for treatment before the scheduled clinical visit and if the participant fulfils the eligibility criteria, they will be invited to participate in the study.

#### **Assignment of interventions: randomization**

#### **Sequence generation {16a}**

After consent, participants are randomly assigned to the study arms with a 1:1 allocation. We will use a simple randomization method with a shuffled deck of sealed envelopes that contain a card with the assigned treatment. The cards are created before the enrollment period and distributed to each of the study sites. No other factors will be taken into consideration for randomization.

#### **Concealment mechanism {16b}**

The envelopes containing the randomization cards are sealed, thus the team member conducting enrollment does not know the content of the envelope.

| 218 | Implementation {16c} |
|---|---|
| 219 | The study staff will ask the participant to select a sealed envelope from the shuffled deck. After |
| 220 | selecting the envelope, the participant will reveal the treatment to themselves and the study staff. |
| 221 | |
| 222 | Assignment of interventions: Blinding |
| 223 | Who will be blinded {17a} |
| 224 | This is an open label clinical trial, while neither the participants nor the study staff will be blinded |
| 225 | to the assigned treatment, staff performing statistical analyses will be masked to treatment |
| 226 | assignment. |
| 227 | Procedure for unblinding if needed {17b} |
| 228 | Not applicable. |
| 229 | Data collection and management |
| 230 | Plans for assessment and collection of outcomes {18a} |
| 231 | A venipuncture blood sample will be collected at 3, 6, and 12 month visits and it will be tested for |
| 232 | RPR titer Study data collected on baseline include basic demographic information, sexual history, |
| 233 | laboratory tests (CD4 count, viral load, RPR titer). On each follow up visit, sexual history, |
| 234 | antibiotic use, symptoms and the RPR titer will be collected. Data will be collected on paper data |
| 235 | collection forms and will be entered into Research Electronic Data Capture (REDCap) (23, 24). |
| 236 | Plans to promote participant retention and complete follow-up {18b} |
| 237 | Study follow-up visits are scheduled to coincide with routine clinic appointments within AHF. |
| 238 | Study staff will send participants a 1 month, 2 week, and 1 day notification prior to their follow-up |
| 239 | appointment. |
| 240 | Data management {19} |

Participant data will be collected on paper data collection forms and entered into RedCap. Data that 241 242 will be entered into RedCap include participant information (name, date of birth, medical record 243 number, contact information) and laboratory results. 244 **Confidentiality {27}** 245 Redcap servers are encrypted, HIPAA-compliant, password protected and accessible only by 246 designated study members. Hard copy data collection forms will be stored into a locked cabinet 247 with limited access only to designated members. 248 249 Plans for collection, laboratory evaluation and storage of biological specimens for genetic or 250 molecular analysis in this trial/future use {33} 251 There are no plans in this trial to evaluate or store biological specimen for genetic or molecular 252 analysis for future use. 253 254 Statistical methods 255 Statistical methods for primary and secondary outcomes {20a} 256 The primary analysis for the main outcome will be conducted on the "Per Protocol" (PP) 257 population. This will include participants who satisfy the inclusion and exclusion criteria, 258 completed treatment (i.e. received the penicillin injection or received all of the cefixime pills), 259 report no adverse events, returned for follow-up visits (3 and/or 6 months) and have an evaluable 260 RPR result. 261 For each treatment group, we will calculate the proportion of PP participants who achieved a 4-fold RPR titer decrease at 3, or 6-months post-treatment and the exact binomial 95% confidence 262 263 interval. 264

| 265 | Interim analyses {21b} |
|---|---|
| 266 | A summary of the enrollment progress, treatment success proportions, adverse events and protocol |
| 267 | deviations will be provided to the Data Safety Monitoring Board members. |
| 268 | |
| 269 | Plans to give access to the full protocol, participant level-data and statistical code {31c} |
| 270 | The protocol of the study is publicly available on clinicaltrials.gov (NCT03660488). Deidentified |
| 271 | data will be available upon request to the study Primary Investigator. |
| 272 | |
| 273 | Oversight and monitoring |
| 274 | Composition of the coordinating center and trial steering committee {5d} |
| 275 | The immediate study research team based in the University of California of Los Angeles meet on a |
| 276 | weekly basis. The immediate team is joined by a wider team of AHF study clinicians, based in |
| 277 | study clinics, who also meet on a weekly basis. |
| 278 | |
| 279 | Composition of the data monitoring committee, its role and reporting structure {21a} |
| 280 | The Data and Safety Monitoring Board (DSMB) will be composed of a physician, biostatistician, |
| 281 | regulatory affairs specialist/ethicist and will oversee the study throughout the 2-year study period. |
| 282 | They will review study activities every 6 months. The committee will review safety data and |
| 283 | clinical efficacy reports and report their decision to the Primary investigator. |
| 284 | |
| 285 | Adverse event reporting and harms {22} |
| 286 | The study site investigators will report serious adverse events and adverse events to the responsible |
| 287 | IRB for that study site in accordance with respective IRB policies and procedures. Follow-up |

288 information to a reported adverse event will be submitted to the IRB as soon as the relevant 289 information is available. 290 291 Frequency and plans for auditing trial conduct {23} 292 The trial and individual clinic sites will be audited at least once during the duration of the study by 293 the study sponsor (AIDS Healthcare Foundation). 294 295 Plans for communicating important protocol amendments to relevant parties (e.g. trial 296 participants, ethical committees) {25} 297 Amendments will be submitted to the IRB according to policies and guidance. Any protocol 298 changes will be promptly communicated to the IRB, the DSMB and the study team. 299 300 **Dissemination plans {31a}** 301 We plan to disseminate study results through peer-reviewed journal publications and conference 302 presentations. Study findings will also be shared with relevant clinical and scientific groups. 303 304 **Discussion** 305 This is a randomized, non-comparative, pilot study evaluating the efficacy of daily oral cefixime 306 400mg for 10 days for the treatment of early syphilis. To our knowledge, this is the first study 307 assessing the efficacy of cefixime for early syphilis. As syphilis rates increase and penicillin 308 shortages continue to occur in the United States and worldwide, alternative treatments that are 309 efficacious for both pregnant and non-pregnant populations, regardless of HIV status are needed (6-8). Already approved and antibiotics in clinical use with favourable pharmacokinetic profile, such 310

311 as cefixime, should be clinically evaluated for alternative treatment options. 312 Data from this pilot study could be used as a foundation to assess the clinical effectiveness for 313 cefixime in early syphilis treatment. Currently, our study is being conducted among non-pregnant 314 individuals. However, subsequent clinical studies should also include women and pregnant women 315 to address the gap in the treatment of maternal syphilis. 316 317 **Trial status** 318 Recruitment was initiated in September 16<sup>th</sup>, 2018 and is currently ongoing. The current protocol 319 version is version 9 (11/20/2020). 320 321 **Declarations** 322 **Authors' contributions {31b}** 323 SM led the writing of the manuscript. CS led the proposal and protocol development and contributed to the writing of the manuscript. DT, PB, CO, and CM contributed to clinical and 324 325 logistical aspects of protocol development. JDK led the proposal and protocol development and 326 developed the treatment algorithm for the protocol. All named authors adhere to the authorship 327 guidelines of Trials. All authors have approved the final manuscript and agreed to publication. 328 329 The database for this study was supported by NIH National Center for Advancing Translational 330 Science (NCATS) UCLA CTSI Grant Number UL1TR001881. 331 Funding {4} 332 The trial is funded by AHF (Grant #20181796). The funding body had no role in the design of the 333 study, collection of data or the writing of this paper, nor will the funding body have a role in 334 analysis, interpretation of data or in writing future manuscripts.

| 335 | |
|---|---|
| 336 | Availability of data and materials {29} |
| 337 | The datasets analyzed during the current study are available from the corresponding author on |
| 338 | reasonable request. |
| 339 | |
| 340 | Ethics approval and consent to participate {24} |
| 341 | The study was approved by Western IRB (IRB# 20181796) and UCLA IRB (IRB# 18-000665). |
| 342 | |
| 343 | Consent for publication {32} |
| 344 | Not applicable |
| 345 | Competing interests {28} |
| 346 | The authors declare that they have no competing interests. |
| 347 | |
| 348 | Author details |
| 349 | 1. Department of Medicine, David Geffen School of Medicine at UCLA, Los Angeles, CA/United |
| 350 | States of America |
| 351 | 2. Department of Medicine, AIDS Healthcare Foundation, Los Angeles, CA/United States of |
| 352 | America |
| 353 | 3. Public Health Division, AIDS Healthcare Foundation, Los Angeles, CA/United States of |
| 354 | America |

#### 355 References

- 356 1. ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine
- 357 (US). Identifier NCT03660488, Cefixime for Alternative Syphilis Treatment; 2018 Sep 6 [cited
- 358 2020 April 29]; Available from: <a href="https://clinicaltrials.gov/ct2/show/NCT03660488">https://clinicaltrials.gov/ct2/show/NCT03660488</a>
- 359 2. Braxton J, Grey J, Harvey A, Kidd S, Presley RJ, Ramirez V, et al. Syphilis surveillance
- 360 supplement 2013–2017 for Sexually transmitted disease surveillance 2017. 2019.
- 361 3. Kojima N, Klausner JDJCer. An update on the global epidemiology of syphilis.
- 362 2018;5(1):24-38.
- World Health Organization. WHO guidelines for the treatment of Treponema pallidum
- 364 (syphilis). 2016
- 365 5. Clement ME, Okeke NL, Hicks CBJJ. Treatment of syphilis: a systematic review.
- 366 2014;312(18):1905-17.
- 367 6. Ghanem KG, Erbelding EJ, Cheng WW, Rompalo AMJCID. Doxycycline compared with
- benzathine penicillin for the treatment of early syphilis. 2006;42(6):e45-e9.
- Wong T, Singh AE, De PJTAjom. Primary syphilis: serological treatment response to
- doxycycline/tetracycline versus benzathine penicillin. 2008;121(10):903-8.
- 371 8. Centers for Disease Control and Prevention. 2015 STD Treatment Guidelines 2015, June 4
- 372 [Available from: <a href="https://www.cdc.gov/std/tg2015/default.htm">https://www.cdc.gov/std/tg2015/default.htm</a>.
- 373 9. Roberts CP, Raich A, Stafylis C, Klausner JDJStd. Alternative Treatments for Syphilis
- 374 During Pregnancy. 2019;46(10):637-40.
- Nurse-Findlay S, Taylor MM, Savage M, Mello MB, Saliyou S, Lavayen M, et al. Shortages
- of benzathine penicillin for prevention of mother-to-child transmission of syphilis: An evaluation
- from multi-country surveys and stakeholder interviews. 2017;14(12).
- 378 11. Taylor MM, Zhang X, Nurse-Findlay S, Hedman L, Kiarie JJBotWHO. The amount of
- penicillin needed to prevent mother-to-child transmission of syphilis. 2016;94(8):559.
- World Health Organization. Shortages of benzathine penicillin. How big is the problem?
- And why it matters 2017 [updated 2017, 27 December
- 382 Available from: https://www.who.int/reproductivehealth/shortages-benzathine-penicillin/en/.
- Liang Z, Chen Y-P, Yang C-S, Guo W, Jiang X-X, Xu X-F, et al. Meta-analysis of
- ceftriaxone compared with penicillin for the treatment of syphilis. 2016;47(1):6-11.
- 385 14. Suprax- Cefixime-Oral Drug Information
- 386 15. Faulkner R, Bohaychuk W, Haynes J, Desjardins R, Yacobi A, Silber BJEjocp. The
- pharmacokinetics of cefixime in the fasted and fed state. 1988;34(5):525-8.
- 388 16. Faulkner R, Fernandez P, Lawrence G, Sia L, Falkowski A, Weiss A, et al. Absolute
- 389 bioavailability of cefixime in man. 1988;28(8):700-6.
- 390 17. Nix DE, Symonds WT, Hyatt JM, Wilton JH, Teal MA, Reidenberg P, et al. Comparative
- 391 pharmacokinetics of oral ceftibuten, cefixime, cefaclor, and cefuroxime axetil in healthy volunteers.
- 392 Pharmacotherapy. 1997;17(1):121-5.
- 393 18. Schatz BS, Karavokiros KT, Taeubel MA, Itokazu GS. Comparison of cefprozil,
- 394 cefpodoxime proxetil, loracarbef, cefixime, and ceftibuten. The Annals of pharmacotherapy.
- 395 1996;30(3):258-68.
- 396 19. Zakeri-Milani P, Valizadeh H, Islambulchilar Z. Comparative bioavailability study of two
- 397 cefixime formulations administered orally in healthy male volunteers. Arzneimittel-Forschung.
- 398 2008;58(2):97-100.
- 399 20. Barbee LA, Nayak SU, Blumer JL, O'Riordan MA, Gray W, Zenilman JM, et al. A Phase 1
- 400 pharmacokinetic and safety study of extended-duration, high-dose cefixime for cephalosporin-
- 401 resistant Neisseria gonorrhoeae in the pharynx. 2018;45(10):677-83.
- 402 21. Rafal'skiĭ V, Kozyrev I, Gustovarova T, Khlybova S, Novoselova A, Filippenko N, et al.
- The efficacy and safety of cefixime and amoxicillin/clavulanate in the treatment of asymptomatic
- bacteriuria in pregnant women: a randomized, prospective, multicenter study. 2013(5):24, 6-8.

- 405 22. Arlington Scientific Inc. RPR card test for syphilis
- 406 2006.
- 407 23. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JGJJobi. Research electronic
- data capture (REDCap)—a metadata-driven methodology and workflow process for providing
- 409 translational research informatics support. 2009;42(2):377-81.
- 410 24. Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, et al. The REDCap
- 411 consortium: Building an international community of software platform partners. 2019;95:103208.